CLINICAL TRIAL: NCT07055841
Title: Single-Arm Exploratory Study of PD-L1 Antibody Plus Neoadjuvant Chemotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiuping Ding (Other)
Responsible Party: Sponsor-Investigator, Xiuping Ding, Dr, Shandong Tumor Hospital
Organization: Shandong Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-OBU-SD-HNC-II-003
Record Dates: First submitted 2025-06-18; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: PD-L1; Local late stage
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — TP protocol; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 (Experimental): TP regimen Adbelimab Surgery or radiotherapy should be performed 1-4 weeks after the completion of neoadjuvant therapy.
  Interventions: Drug: Adebrelimab; Drug: TP regimen; Procedure: Surgery or radiotherapy

INTERVENTIONS:
Drug: Adebrelimab — 1200mg, intravenous infusion, D1， Every three weeks, there are two cycles in total.
Drug: TP regimen — TP regimen: Docetaxel 75 mg/m2, intravenous infusion, D1， Cisplatin 75 mg/m2, intravenous infusion, D1， Every three weeks, there are two cycles in total.
Procedure: Surgery or radiotherapy — Surgery or radiotherapy should be performed 1-4 weeks after the completion of neoadjuvant therapy.

SUMMARY:
This single-arm exploratory study plans to enroll 69 locally advanced head and neck squamous cell carcinoma (LA-HNSCC) patients. Participants will receive Adebrelimab (PD-L1 antibody) plus TP regimen (docetaxel/cisplatin) as neoadjuvant therapy for 1-4 weeks, followed by surgery and subsequent follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with head and neck squamous cell carcinoma diagnosed by histology or cytology;
* 2. Have not received systematic treatment for head and neck squamous cell carcinoma in the past;
* 3. According to the AJCC TNM staging system, it is divided into stages III-IVB;
* 4. ECOG score: 0-1 point;
* 5. Expected survival period ≥ 12 weeks;
* 6. The main organ functions well and the laboratory test data meets the following standards: (1) Blood routine: absolute neutrophil count ≥ 1.5 × 109/L (or greater than the lower limit of normal laboratory values in the research center), platelet count ≥ 100 × 109/L, hemoglobin ≥ 90g/L; (2) Liver function: serum total bilirubin ≤ 1.5 times the upper limit of the standard value (ULN), AST and ALT ≤ 2.5 times ULN. If the patient has liver metastasis, this standard is ≤ 5 times ULN; (3) Renal function: CrCl ≥ 60 ml/min/1.73 m2 (calculated according to the Cockcroft Gault formula);
* 7. Female subjects with fertility, as well as male subjects with partners who are fertility women, are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period, at least 6 months after the last use of adebelimab, and at least 6 months after the last use of chemotherapy;
* 8. Voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* 1. There is uncontrollable pleural effusion, pericardial effusion, or peritoneal effusion that requires repeated drainage;
* 2. Have a history of allergies to any components of Adabelimab in the past;
* 3. Have received any of the following treatments:

  1. Received any other investigational drug within 4 weeks prior to the first use of the investigational drug or had a half-life of no more than 5 from the last investigational drug;
  2. Simultaneously enrolled in another clinical study, unless it is an observational (non interventional) clinical study or an interventional clinical study follow-up;
  3. Received anti-tumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, or tumor embolization) within 2 weeks prior to the first use of the investigational drug;
  4. Subjects who need to receive corticosteroids (equivalent to>10mg prednisone per day) within 2 weeks prior to the first use of the study drug. Allow the use of hormones for routine chemotherapy pretreatment without the need for dose adjustment. Other special circumstances require communication with the researcher. In the absence of active autoimmune diseases, inhalation or local use of steroids and corticosteroids with a dosage greater than 10mg/day of prednisone efficacy dose are allowed as substitutes for adrenal cortex hormones;
  5. Individuals who have received anti-tumor vaccines or have received live vaccines within 4 weeks prior to the first administration of the study drug;
  6. Having undergone major surgery or suffered severe trauma within 4 weeks prior to the first use of the investigational drug;
  7. Patients who have received previous treatment with paclitaxel drugs;
* 4. The toxicity of previous anti-tumor treatments has not recovered to ≤ CTCAE 5.0 Grade 1 (excluding hair loss) or the level specified in the inclusion/exclusion criteria;
* 5. Active autoimmune diseases, history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to the above diseases or syndromes); Excluding childhood asthma/allergies with vitiligo or those who have already recovered, patients who do not require any intervention in adulthood; Autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with a stable dose of insulin;
* 6. Have a history of immune deficiency, including HIV test positive, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation, or active hepatitis (hepatitis B reference: HBV DNA test value exceeds 500 IU/ml or 2500 copies/mL);
* 7. The subject has uncontrolled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year; (4) Clinically significant supraventricular or ventricular arrhythmias that have not been clinically intervened or are still poorly controlled after clinical intervention;
* 8.Within 4 weeks prior to the first use of the investigational drug, there has been a severe infection (CTCAE 5.0>grade 2), such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc; Baseline chest imaging examination suggests the presence of active pulmonary inflammation, symptoms and signs of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous administration Or intravenous use of antibiotics for treatment, except for prophylactic use of antibiotics;
* 9. History of interstitial lung disease (excluding history of radiation pneumonia and non infectious pneumonia that have not been treated with steroids);
* 10. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within the past year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than one year ago but without formal treatment;
* 11. Diagnosed with any other malignant tumor within 5 years prior to the first use of the investigational drug, except for malignant tumors with low-risk metastasis and mortality risk (5-year survival rate>90%), such as basal cell or squamous cell carcinoma or cervical carcinoma in situ that have been adequately treated;
* 12. Pregnant or lactating women;
* 13. According to the researcher's assessment, there may be other factors that could force the subject to terminate the study midway, such as suffering from other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of trial data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment to first efficacy evaluation (around 6-8 weeks)
  Objective response rate (ORR)

SECONDARY OUTCOMES:
pCR | Evaluate based on pathological results, with an evaluation period from enrollment to 2 weeks after surgery
  pathological complete response，pCR
R0 resection rate | Evaluate based on pathological results, with an evaluation period from enrollment to 2 weeks after surgery
  R0 is the ratio of no residual material under the microscope after resection.
EFS | The time from enrollment to the first occurrence of endpoint events such as disease progression and death(maximum follow-up time of 2 years)
  Event-Free Survival（EFS）
Adverse event incidence rate | Follow up from enrollment until 90 days after the last treatment
  Adverse events that occurred during the research process

CONTACTS AND LOCATIONS:
Overall Officials: wanjun chen, physician, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No